CLINICAL TRIAL: NCT01854411
Title: Ibuprofen and Ketoprofen Concentrations in Human Mature Milk. PK Study in Breastmilk AOR-10127 "Antalait" Study
Brief Title: Study of Analgesics Drug and Human Milk Transfer in Mature Milk, to Avoid Breastfeeding Cessation Without Scientific Probes
Acronym: ANTALAIT
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI09048; AOR10127
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Analgesics Use During Breastfeeding and Concentrations in Human Mature Milk
Keywords: Analgesics; Ibuprofene; Ketoprofene; Breastmilk; Relative Infant Dose; Theoric Infant Dose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — human breast milk
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- analgesic dose measure: breastfeeding mother who will take analgesics
  Interventions: Other: analgesic measure

INTERVENTIONS:
Other: analgesic measure — ibuprofen and ketoprofen measured into breast milk

SUMMARY:
The purpose of this study is to determine whether ibuprofen and ketoprofen do not enter into mature breastmilk that could allowed breastfeeding during a long time

DETAILED DESCRIPTION:
Analgesics are frequently used to prevent and treat pain and inflammatory disease.

Due to a lack of information on drug's human milk transfer, breastfeeding is sometimes contraindicated. Mothers are advised to either stop breastfeeding or if they don't, not to treat themselves. Since the fatal neonatal case with codeine during breastfeeding, analgesics are being reviewed. Ibuprofen seems to have the best benefit-risk ratio during the post-partum period. However there are no pharmacologic data about the use of ibuprofen during breastfeeding, after the colostrum phase.

This study aims to determine the relative infant dose (RID) of ibuprofen in human mature milk. Considering the increased interest in NSAIDs in light of the codeine case, this is an important information. It will help health practitioners when advising and treating breastfeeding women.

ELIGIBILITY:
Inclusion Criteria:

* breastfeeding women after the first week of delivery
* breastfeeding women treated by ketoprofen or ibuprofen per os more than 24 hours
* Written Informed Consent

Exclusion Criteria:

* breastfeeding women treated by naproxene
* Curator or justice decision's

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Lactarium, Maternal care, Consultant of Lactation
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-09; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
concentration of ibuprofene in human mature milk. | 6 months
concentration of ketoprofene in human mature milk | 6 months

SECONDARY OUTCOMES:
comparison between ibuprofene and ketoprofene concentrations in the human breastmilk | 6 months
  To compare the concentrations of ibuprofene and ketoprofene in the human breastmilk in correlation with the maturity

CONTACTS AND LOCATIONS:
Overall Officials: virginie rigourd, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- hopital Saint Antoire, Paris, France

REFERENCES:
- See also: Medic-Al network to help the women and investigators to receive specialize information's about breastfeeding and medications — http://reseau-medic-al.fr/index.php